CLINICAL TRIAL: NCT00445978
Title: A Phase 2a, Multicenter, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, and Efficacy of 6R-BH4 in Subjects With Sickle Cell Disease
Brief Title: A Phase 2 Study of the Effects of 6R-BH4 in Subjects With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCD-001
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; SCD; 6R-BH4; BH4; sapropterin dihydrochloride; endothelial dysfunction; Nitric Oxide; NO
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sapropterin dihydrochloride (Experimental): 2.5, 5, 10, 20 mg/kg/day of sapropterin dihydrochloride during a 16-week dose escalation phase, with dose levels increasing within subjects every 4 weeks, with an optional extension phase at the highest tolerated dose for up to a total of 2 years.
  Interventions: Drug: Sapropterin Dihydrochloride

INTERVENTIONS:
Drug: Sapropterin Dihydrochloride — Subjects will receive oral, once-daily (for 2.5, 5, 10mg/kg/day doses) or twice-daily (for the 20 mg/kg/day dose) sapropterin dihydrochloride during a 16-week dose escalation phase, with dose levels increasing within subjects every 4 weeks as follows: 2.5, 5, 10, and 20 mg/kg/day. Dosing was with 100 mg tablets and rounded to the nearest whole tablet. Each dose was taken within 1 hour after the morning meal. Subjects may continue in an optional extension phase at the highest tolerated dose for up to a total of 2 years.
  Other Names: 6R-BH4

SUMMARY:
This Phase 2a, multicenter, open-label, dose-escalation study is designed to assess the safety and biologic activity of daily oral administration of 4 escalating doses of sapropterin dihydrochloride over 16 weeks in subjects with sickle cell disease. During an optional extension phase, the study will assess the safety, tolerability, and efficacy of extended treatment with sapropterin dihydrochloride, for a total of up to 2 years; The extension phase of this study was terminated.

DETAILED DESCRIPTION:
This Phase 2a, multicenter, open-label, dose-escalation study was designed to assess the safety and biological activity of once-daily (or twice-daily [BID], only for the highest dose level) oral administration of 4 escalating doses of sapropterin dihydrochloride to subjects with Sickle Cell Disease (SCD); 32 subjects were enrolled in the dose-escalation phase of this study. Subjects received oral, once daily (for 2.5, 5, and 10 mg/kg/day) or BID (for 20 mg/kg/day) doses of sapropterin dihydrochloride during a 16-week, dose-escalation period, with dose levels increasing within subjects every 4 weeks, as follows: 2.5, 5, 10, and 20 mg/kg/day. At the highest dose level (20 mg/kg/day), the total dose of sapropterin dihydrochloride was divided, half of the tablets taken in the morning within 1 hour after a meal, and half approximately 12 hours later (or BID) within 1 hour after a meal. The extension phase of this study was terminated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD, as confirmed by hemoglobin electrophoresis.
* At least 15 years of age.
* Dosage of medication(s) used to treat cardiac disease, hypertension (eg, calcium-channel blockers), elevated cholesterol, iron overload (eg, desferoxamine) and type 2 diabetes must be unchanged for at least 30 days prior to Screening.
* Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Willing and able to comply with all study procedures.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been menopausal for at least 2 years, or had a tubal ligation at least 1 year prior to Screening, or who have had a total hysterectomy.

Exclusion Criteria:

* Requires chronic hypertransfusion therapy.
* Sickle cell crisis during the 30 days prior to Screening.
* Myocardial infarction, cerebral vascular accident, or pulmonary embolism during the 6 months prior to Screening.
* History of bone marrow or hematopoietic stem cell transplantation.
* Hepatic dysfunction (alanine aminotransferase [ALT][SGPT] > 2 times the upper limit of normal [ULN]).
* Renal dysfunction with serum creatinine > 1.5 mg/dL.
* On outpatient oxygen therapy, or continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BiPAP) therapy.
* Uncontrolled hypertension (defined as blood pressure > 135/85 mm Hg) at Screening.
* History of chronic symptomatic hypotension.
* Concurrent disease or condition that would interfere with study participation or safety, including, but not limited to: bleeding disorders, history of syncope or vertigo, severe gastroesophageal reflux disease (GERD), arrhythmia, organ transplant, organ failure, type 1 diabetes mellitus (subjects with type 2 diabetes are allowed), or serious neurological disorders (including seizures).
* Hydroxyurea therapy during the 3 months prior to Screening or anticipated need for hydroxyurea during the course of the study.
* Treatment with any phosphodiesterase (PDE) 5 inhibitor (Viagra®, Cialis®, Levitra® or Revatio™), any PDE 3 inhibitor (eg, cilostazol, milrinone, or vesnarinone), pentoxifylline (Trental®), nitrate/nitrite-based vasodilators, bosentan (Tracleer®), L-arginine, levodopa, or dietary supplements containing L-arginine or gingko biloba within 30 days prior to Screening, or anticipated need for treatment with any of these agents during the course of the study.
* Requirement for concomitant treatment with any drug known to inhibit folate metabolism (eg, methotrexate).
* Previous treatment with vascular endothelial growth factor (VEGF) or VEGF inhibitors.
* Has known hypersensitivity to sapropterin dihydrochloride or its excipients.
* Use of any investigational product, device, or any formulation of BH4 within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Any condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saba Sile, MD, Study Director — BioMarin Pharmaceutical
Locations (12):
- United States (12):
  - Washington D.C., District of Columbia
  - Augusta, Georgia
  - Savannah, Georgia
  - Indianapolis, Indiana
  - Detroit, Michigan
  - Flint, Michigan
  - Hackensack, New Jersey
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Galveston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia

REFERENCES:
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter dose escalation study with 12 sites in the US in subjects with sickle cell disease (SCD). Only subjects with HbSS (homozygous SCD) and HbSC (heterozygous SCD) genotypes and at least 15 years of age were enrolled.
Pre-assignment Details: Dose escalation was to take place at Week 4, 8, and 12; however some subjects initially maintained the previous dose and received escalated doses at a later time point during the dose interval. This delay was to adhere to the study protocol for escalation (for example, if a subject missed the appointment for PAT testing, dose escalation was delayed until testing could be performed), not due to safety concerns. Subjects not escalated in dose either maintained or reduced dose.
Groups:
- Sapropterin Dihydrochloride: Sapropterin dihydrochloride: Subjects will receive oral tablets, once-daily (for 2.5, 5, 10mg/kg/day doses) or twice-daily (for the 20 mg/kg/day dose) of sapropterin dihydrochloride during a 16-week dose escalation phase, with dose levels increasing within subjects every 4 weeks as follows: 2.5, 5, 10, and 20 mg/kg/day. Prior to dose escalation, the investigator evaluated each subject's safety profile at the previous dose level to determine if the subject would escalate to the next dose level; maintain the same dose; or de-escalate to the previous dose.
Period: Week 0 - Week 4 (2.5 mg/kg/Day)
Arm/Group | Sapropterin Dihydrochloride
Started | 32
Completed | 29
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Study Compliance | 1
Period: Week 4 - Week 8 (5 mg/kg/Day)
Arm/Group | Sapropterin Dihydrochloride
Started | 29
Received Escalated Dose | 29
Completed | 25
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrew Consent | 1
Period: Week 8 - Week 12 (10 mg/kg/Day)
Arm/Group | Sapropterin Dihydrochloride
Started | 25
Received Escalated Dose | 25
Completed | 24
Not Completed | 1
Not completed — Pregnancy | 1
Period: Week 12 - Week 16 (20 mg/kg/Day)
Arm/Group | Sapropterin Dihydrochloride
Started | 24
Received Escalated Dose | 21
Completed | 23
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All Treated Subjects
Groups:
- Sapropterin Dihydrochloride: Sapropterin dihydrochloride: Subjects will receive oral tablets, once-daily (for 2.5, 5, 10mg/kg/day doses) or twice-daily (for the 20 mg/kg/day dose) of sapropterin dihydrochloride during a 16-week dose escalation phase, with dose levels increasing within subjects every 4 weeks as follows: 2.5, 5, 10, and 20 mg/kg/day.
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 32
SCD Genotype [Number; unit: participants]
  SS (homozygous, 2 hemoglobin S alleles) | 19
  SC (heterozygous, 1 hemoglobin S allele, 1 hemoglobin C allele) | 13
PAT (peripheral arterial tonometry) at baseline (Ratio) [Count of Participants; unit: Participants] — PAT serves as a surrogate to assess endothelial function and arterial stiffness.
  Participants
    Normal (PAT > 1.67) | 9
    Abnormal (PAT</= 1.67) | 18
    Missing | 5
TRV (tricuspid regurgitant velocity) at baseline (m/sec) [Count of Participants; unit: Participants] — TRV >/= 2.5 m/sec indicates the presence of pulmonary hypertension.
  Participants
    TRV< 2.5 | 18
    TRV>/= 2.5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse events (TEAE) is any adverse events that newly appeared, increased in frequency or worsened in severity following initiation of study drug administration.
Time Frame: Up to 16 weeks
Population: All Treated Subjects
Measure: Count of Participants; unit: Participants
Groups:
- Sapropterin Dihydrochloride 2.5 mg/kg/Day: Sapropterin dihydrochloride 2.5 mg/kg/day at Incidence
- Sapropterin Dihydrochloride 5.0 mg/kg/Day: Sapropterin dihydrochloride 5.0 mg/kg/day at Incidence
- Sapropterin Dihydrochloride 10.0 mg/kg/Day: Sapropterin dihydrochloride 10.0 mg/kg/day at Incidence
- Sapropterin Dihydrochloride 20.0 mg/kg/Day: Sapropterin dihydrochloride 20.0 mg/kg/day at Incidence
Arm/Group | Sapropterin Dihydrochloride 2.5 mg/kg/Day | Sapropterin Dihydrochloride 5.0 mg/kg/Day | Sapropterin Dihydrochloride 10.0 mg/kg/Day | Sapropterin Dihydrochloride 20.0 mg/kg/Day
Number analyzed (Participants) | 32 | 29 | 25 | 21
Participants
  Subjects with any adverse event | 27 | 18 | 20 | 15
  Subjects with any serious adverse events | 3 | 2 | 6 | 3
  Subjects with any treatment-related adverse event | 9 | 4 | 6 | 3
  Any subject with a treatment-related serious adverse event | 0 | 1 | 2 | 0
  Any subject with an AE causing study discontinuation | 1 | 1 | 0 | 1
  Any subject with an SAE causing study discontinuation | 1 | 1 | 0 | 0
  Death | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in the Peripheral Arterial Tonometry (PAT) Scores
Description: The PAT score was calculated using the ratio between the arterial pulse wave amplitude following a 5-minute arterial occlusion in the forearm to the pre-occlusion value (Reactive Hyperemia Index). A value of </= 1.67 represents an impaired response or endothelial dysfunction. Change in PAT from Baseline to posttreatment visit is calculated by subtracting the Baseline measurement from the posttreatment measurement.
Time Frame: At Baseline, Week 4, 8, 12 and 16.
Population: At each timepoint of the dose-escalation phase, subjects with evaluable PAT score at the corresponding timepoint and baseline were included in the change from baseline analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 27
Ratio
  Baseline | 1.5815 (0.4292)
  Change from Baseline to Week 4: number analyzed (Participants) | 22
  Change from Baseline to Week 4 | 0.1317 (0.4811)
  Change from Baseline to Week 8: number analyzed (Participants) | 21
  Change from Baseline to Week 8 | 0.2852 (0.6020)
  Change from Baseline to Week 12: number analyzed (Participants) | 22
  Change from Baseline to Week 12 | 0.3656 (0.5004)
  Change from Baseline to Week 16: number analyzed (Participants) | 21
  Change from Baseline to Week 16 | 0.3604 (0.8800)

3. Secondary Outcome: Change From Baseline in the Urine 8-Isoprostane
Description: Change in urine 8-isoprostane from Baseline to post-treatment visit is calculated by subtracting the Baseline measurement from the post-treatment measurement. This outcome was used to assess change in oxidative stress.
Time Frame: At Baseline, Week 4, 8, 12 and 16.
Population: At each timepoint of the dose-escalation phase, subjects with urine 8-isoprostane at the corresponding timepoint and baseline were included in the change from baseline analysis.
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 32
pg/mg creatinine
  Baseline | 1019.68 (479.90)
  Change from Baseline to Week 4: number analyzed (Participants) | 29
  Change from Baseline to Week 4 | -27.58 (622.53)
  Change from Baseline to Week 8: number analyzed (Participants) | 24
  Change from Baseline to Week 8 | -69.75 (402.83)
  Change from Baseline to Week 12: number analyzed (Participants) | 23
  Change from Baseline to Week 12 | 24.71 (355.71)
  Change from Baseline to Week 16: number analyzed (Participants) | 22
  Change from Baseline to Week 16 | -275.19 (566.99)

4. Secondary Outcome: Change From Baseline in the Urine Spot Albumin to Creatinine Ratio
Description: Change in Urine Albumin to Creatinine Ratio from Baseline to post-treatment visit is calculated by subtracting the Baseline measurement from the post-treatment measurement. This outcome was used to assess change in renal function.
Time Frame: At Baseline, Week 4, 8, 12 and 16.
Population: At each timepoint of the dose-escalation phase, subjects with urinary spot albumin to creatinine at the corresponding timepoint and baseline were included in the change from baseline analysis.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 26
mg/mmol
  Baseline | 17.88 (42.44)
  Change from Baseline to Week 4: number analyzed (Participants) | 18
  Change from Baseline to Week 4 | 1.66 (27.43)
  Change from Baseline to Week 8: number analyzed (Participants) | 16
  Change from Baseline to Week 8 | -5.51 (25.31)
  Change from Baseline to Week 12: number analyzed (Participants) | 14
  Change from Baseline to Week 12 | -10.76 (24.73)
  Change from Baseline to Week 16: number analyzed (Participants) | 15
  Change from Baseline to Week 16 | -9.32 (23.82)

5. Secondary Outcome: Change From Baseline in the Tricuspid Regurgitant Velocity (TRV)
Description: Change in tricuspid regurgitant velocity (TRV) from Baseline to post-treatment visit is calculated by subtracting the Baseline measurement from the post-treatment measurement.
Time Frame: At Baseline, Week 4, 8, 12 and 16.
Population: At each timepoint of the dose-escalation phase, subjects with tricuspid regurgitant velocity at the corresponding timepoint and baseline were included in the change from baseline analysis.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 32
m/sec
  Baseline | 2.09 (0.84)
  Change from Baseline to Week 4: number analyzed (Participants) | 27
  Change from Baseline to Week 4 | 0.09 (0.53)
  Change from Baseline to Week 8: number analyzed (Participants) | 25
  Change from Baseline to Week 8 | 0.03 (0.73)
  Change from Baseline to Week 12: number analyzed (Participants) | 23
  Change from Baseline to Week 12 | 0.01 (0.43)
  Change from Baseline to Week 16: number analyzed (Participants) | 22
  Change from Baseline to Week 16 | 0.16 (0.72)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Sapropterin Dihydrochloride 2.5 mg/kg/Day | Sapropterin Dihydrochloride 5.0 mg/kg/Day | Sapropterin Dihydrochloride 10.0 mg/kg/Day | Sapropterin Dihydrochloride 20.0 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29 | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/32 | 2/29 | 6/25 | 3/21
Other Adverse Events (participants affected / at risk) | 27/32 | 18/29 | 20/25 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin Dihydrochloride 2.5 mg/kg/Day (N=32) | Sapropterin Dihydrochloride 5.0 mg/kg/Day (N=29) | Sapropterin Dihydrochloride 10.0 mg/kg/Day (N=25) | Sapropterin Dihydrochloride 20.0 mg/kg/Day (N=21)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 3 | 2 | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin Dihydrochloride 2.5 mg/kg/Day (N=32) | Sapropterin Dihydrochloride 5.0 mg/kg/Day (N=29) | Sapropterin Dihydrochloride 10.0 mg/kg/Day (N=25) | Sapropterin Dihydrochloride 20.0 mg/kg/Day (N=21)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 9 | 7 | 10 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 2 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 4 | 1 | 2 | 0
Insomnia (Nervous system disorders) | 1 | 0 | 2 | 1
Migraine (Nervous system disorders) | 2 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Flank pain (General disorders) | 0 | 1 | 0 | 0
Oedma (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Allergic Sinusitis (Immune system disorders) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Vaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Tenderness (General disorders) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroenteritis viral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin papilloma (Infections and infestations) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint sprain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Albumin urine (Investigations) | 1 | 0 | 0 | 0
Albumin urine present (Investigations) | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 1 | 0 | 0
Cardiac mumur (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Mammogram abnormal (Investigations) | 0 | 0 | 1 | 0
Urinary sediment present (Investigations) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Ecchymosis (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The quality of the sickle cell crisis data collected was not adequate to make any conclusions about sapropterin dihydrochloride and sickle cell painful or vaso-occlusive crisis due to selection and reporting bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days